CLINICAL TRIAL: NCT05032092
Title: Evaluation of Efficacy of Comprehensive Genomic Tumour Profiling (CGP) From Liquid and/or Tissue Biopsy in Patients With Locally Advanced and/or Metastatic Solid Cancer
Acronym: SOUND
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1168/2021
Record Dates: First submitted 2021-08-19; First posted 2021-09-02 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Carcinoma; Metastatic Cancer
Keywords: Comprehensive Genomic Tumour Profiling; Targeted Therapy; Progression Free Survival; Next Generation Sequencing; Molecular Tumour Board; Tumour-specific Therapy
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Open, Prospective, Multicentre IVD (in vitro diagnostic device) Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients with locally advanced and/or metastasized solid cancer (Experimental): Liquid biopsies of all 235 study patients will be analysed with FoundationOne®Liquid CDx.
  Tissue biopsies from all study patients for whom a tissue biopsy is available will be analysed with FoundationOne® CDx and IHC (approximately 50% of the enrolled patients).
  Biomarker Monitoring of study patients receiving matched therapy with AVENIO ctDNA Expanded Kit.
  Interventions: Diagnostic Test: Next Generation Sequencing; Genetic: Biomarker Monitoring

INTERVENTIONS:
Diagnostic Test: Next Generation Sequencing — Molecular analysis of liquid biopsy.
  Other Names: FoundationOne®Liquid CDx
Diagnostic Test: Next Generation Sequencing — Molecular analysis of tissue biopsy.
  Other Names: FoundationOne® CDx
Genetic: Biomarker Monitoring — Biomarker Monitoring of study patients receiving matched therapy.
  Other Names: AVENIO ctDNA Expanded Kit

SUMMARY:
The aims of this study are

* to evaluate the efficacy of comprehensive genomic tumour profiling (CGP) from liquid and/or tissue biopsy in patients with locally advanced and/or metastatic solid cancer.
* to evaluate and describe the impact of treatment decisions based on CGP on individual progression free survival in patients with locally advanced and/or metastatic solid cancer
* to evaluate and describe similarities and differences between the treatment suggestions based on CGP/IHC (immuno-histochemistry) of tissue biopsy and liquid biopsy.

In patients with locally advanced and/or metastatic carcinoma the primary efficacy objective of the study is, to observe and describe the PFS (progression-free survival) of the matched treatment compared to the PFS of the most recent therapy.

DETAILED DESCRIPTION:
The SOUND study will be exploring the treatment rates and outcomes of CGP-driven targeted treatment in patients with advanced or metastasized cancer. It will use a substantially larger gene-panel than previous studies in Austria. Departing from the routine clinical practice, study patients will have the opportunity to have CGP from liquid and/or tissue biopsy. The treatment decision will be discussed within a molecular tumour board consisting of experts in clinical oncology, human genetics and pathology. The treatment decision process will be supported and documented by a software.

Data from the SOUND study will cover the whole analysis process, the reasons for the treatment decision, reasons for getting or not-getting a matched treatment as well as the outcome, treatment and hospitalisation costs. The SOUND study will give valuable insights into the clinical practice of CGP-driven therapy in Austria and describe the experience and the possible restrictions. Considering the differing conditions in Austria, the SOUND study will generate data that might be useful for best practice sharing with other countries in the future.

ELIGIBILITY:
Inclusion Criteria:

* Initial diagnosis of histologically confirmed locally advanced and/or metastatic solid cancer
* Radiologically confirmed progression under the most recent therapy
* No further evidence-based drug treatment is established, or no satisfactory alternative treatments are available for the locally advanced and/or metastasized carcinoma
* Further therapy is medically feasible
* ECOG (Eastern Cooperative Oncology Group) performance status 0-2
* Life expectancy of at least 12 weeks
* Written informed consent and willingness to cooperate during the course of the study
* Capability to understand the intention and the consequences of the study

Exclusion Criteria:

* Untreated CNS (central nervous system) metastases. Patients with treated CNS metastases are eligible if they are clinically stable with regard to neurologic function
* Pregnant or breast feeding
* Other malignomas, diagnosed < 5a before inclusion (except localized squamous cell carcinomas of the skin, surgically curable melanomas of the skin, basal cell carcinomas of the skin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Estimated)
Dates: Start 2021-11-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Progression Free Survival (PFS): (matched therapy) /PFS (most recent therapy) > 1.3 | Start of treatment to radiomorphologically confirmed progression of disease, that is on average about 4 months
  To observe and describe the PFS of the matched treatment compared to the PFS of the most recent therapy, PFS = number of calendar days from start treatment to progression of disease

SECONDARY OUTCOMES:
Number of potentially actionable targets | Within seven days after NGS report at Molecular Tumour Board, i.e. 14 to 30 days after enrolment of patient
  To evaluate the number of targets identified with NGS (next-generation sequencing) and IHC, that are potentially actionable with an approved drug on-label, off-label or an experimental drug per patient
Proportion of patients with potentially actionable targets | A maximum of 30 months after first patient first visit
  To investigate the proportion of patients with targets actionable by an approved drug on-label, off-label or an experimental drug.
Calendar days from enrolment into the study to the date of death or last visit alive | Enrolment to death or last visit alive, that is on average about 8 months
  To observe and describe overall survival (OS)
Proportion of patients with best overall response of either complete response (CR) or partial response (PR), based on their overall response | A maximum of 30 months after first patient first visit
  To observe and describe objective response rate (ORR), Response will be evaluated by the investigator as defined by RECIST 1. or irRECIST
Proportion of patients with successful molecular profiling from liquid or tissue biopsy, in whom a matched therapy was recommended | A maximum of 30 months after first patient first visit
  To investigate the proportion of patients with successful molecular profiling

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Jost, Univ.Prof.Dr.MD,, Principal Investigator — Medical University of Graz, Department of Internal Medicine, Division of Clinical Oncology; Armin Gerger, Univ.Prof.,MD., Principal Investigator — Medical University of Graz, Department of Internal Medicine, Division of Clinical Oncology
Locations (6):
- Austria (6):
  - University Hospital Salzburg, Department of Internal Medicine III, Salzburg, Salzburg
  - Medical University of Innsbruck, Department of Hematology and Oncology, Innsbruck, Tyrol
  - Ordensklinikum Linz, Linz, Upper Austria
  - Landeskrankenhaus Feldkirch, Department of Internal Medicine II, Feldkirch, Vorarlberg
  - Landesklinikum Amstetten, Amstetten
  - Medical University of Graz, Graz

IPD SHARING:
Plan to Share IPD: No